CLINICAL TRIAL: NCT05145205
Title: Effect of Laparoscopic Sleeve Gastrectomy vs Laparoscopic Roux-en-Y Gastric Bypass on Weight Loss in Patients With Morbid Obesity
Brief Title: Laparoscopic Sleeve Gastrectomy vs Laparoscopic Roux-en-Y Gastric Bypass
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdulkarim Hasan, Researcher, Al-Azhar University
Other Study IDs: AUH210021
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Laparoscopic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LSG
  Interventions: Procedure: Sleeve gastrectomy
- RYGB
  Interventions: Procedure: Laparoscopic Roux-en-Y gastric bypass

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Bougie was applied over the lower curvature to adjust the gastric tube then longitudinal amputation of the stomach was performed for about 4 to 6 cm per pecker of the pylorus to the corner of His. No supportive materials were used, and over-suturing of the basic line performed only over the points of bleeding.
  All resected specimens were sent to histopathology laboratory for examination.
  Groups: LSG
Procedure: Laparoscopic Roux-en-Y gastric bypass — An antecolic and antegastric RYGB become executed with a 150 cm alimentary limb with both a linearly or circularly kink (25 mm) gastrojejunostomy in step with the desire of the surgeon. A 50-cm-lengthy biliopancreati
  Groups: RYGB

SUMMARY:
This is a retrospective work on 200 morbid obese patients randomized and categorized into 2 groups according to the treatment method: the laparoscopic sleeve gastrectomy (LSG) and LRYGB groups, within the period from 2014 to 2019 and matched weight dissipation, complications, life quality, and negative events

ELIGIBILITY:
Inclusion Criteria:

* All patients of (Body Mass Index) more than 40, with at least 1 comorbidity

Exclusion Criteria:

* All patients of (Body Mass Index) less than 40,
* No comorbidities
* Patients who refused the surgical procedures.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study included Egyptian patients with age ranging from 18 to 70 seeking surgical operation for obesity.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
weight dissipation | 12 months
  decrease the body mass index by 1 or more

CONTACTS AND LOCATIONS:
Locations (1):
- Azhar faculty of medicine, Cairo, Egypt